CLINICAL TRIAL: NCT07046923
Title: A First-in-Human, Phase 1a/1b Trial to Assess the Safety, Tolerability and Preliminary Efficacy of LY4175408, an Antibody Drug Conjugate Targeting Protein Tyrosine Kinase 7-Expressing Tumor Cells, in Participants With Selected Advanced Solid Tumors
Brief Title: A Study of LY4175408 in Participants With Advanced Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 27401; J6D-MC-JSDA (Other: Eli Lilly and Company); 2025-521916-20-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Endometrial Neoplasms; Neoplasm Metastasis; Triple Negative Breast Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Endometrial Neoplasms; Neoplasm Metastasis; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1a Dose Escalation (Cohort A1) (Experimental): Escalating doses of LY4175408 administered intravenously (IV)
  Interventions: Drug: LY4175408
- Phase 1a Dose Optimization (Cohort A2) (Experimental): Two or more doses of LY4175408 (evaluated during dose escalation) administered IV
  Interventions: Drug: LY4175408
- Phase 1b Dose Expansion (Cohort B) (Experimental): LY4175408 administered IV
  Interventions: Drug: LY4175408

INTERVENTIONS:
Drug: LY4175408 — IV infusion

SUMMARY:
The purpose of this study is to measure the safety and efficacy of LY4175408 in participants with selected advanced cancer. In addition, this study will evaluate how much LY4175408 gets into the bloodstream, how it is broken down, and how long it takes the body to get rid of it. Participation could last up to 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Have one of the following advanced or metastatic solid tumor cancers:

  * Non-small cell lung cancer (NSCLC)
  * Small cell lung cancer (SCLC)
  * Endometrial cancer
  * Triple negative breast cancer (TNBC) (characterized by HR-negative disease and HER2-negative expression according to American Society of Clinical Oncology (ASCO) - College of American Pathologists guidelines).
* Received all standard therapies for which the individual was deemed to be an appropriate candidate by the treating investigator; OR the individual is refusing the remaining most appropriate standard of care treatment; OR there is no standard therapy available for the disease.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤1.
* For dose optimization/dose and expansion cohorts (Cohort A2, Cohort B): Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

Exclusion Criteria:

* Prior treatment with a protein tyrosine kinase 7 (PTK7) antibody-drug conjugate (ADC) with a topoisomerase I inhibitor as payload (prior therapy with a PTK7 ADC with a non-topoisomerase I inhibitor payload OR non-PTK7 ADC with any payload is permitted).
* Any serious unresolved toxicities from prior therapy.
* Individual with known or suspected history of uncontrolled central nervous system (CNS) metastases.
* Individual with active uncontrolled systemic bacterial, viral, fungal, or parasitic infection.
* Significant cardiovascular disease.
* Prolongation of QT interval corrected for heart rate using Fridericia's formula (QTcF) > 470 milliseconds (ms)
* History of pneumonitis/interstitial lung disease.
* Individuals who are pregnant, breastfeeding, or plan to breastfeed during the trial or within 30 days of the last dose of trial intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Phase 1a-Number of Participants with Dose Limiting Toxicities of LY4175408 | 1 Cycle (21 days)
Phase 1b-Overall Response Rate (ORR): Percentage of Participants with Best Response of Complete Response (CR) or Partial Response (PR) | Baseline up to approximately 4 years
  Per investigator assessed Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)

SECONDARY OUTCOMES:
Phase 1a and 1b-Pharmacokinetics (PK): Minimum Plasma Concentration (Cmin) of LY4175408 (total antibody, conjugated antibody, free payload) | First 4 cycles (84 days)
Phase 1a and 1b-PK: Area under the Concentration versus Time Curve (AUC) of LY4175408 (total antibody, conjugated antibody, free payload) | First 4 cycles (84 days)
Phase 1a-ORR: Percentage of Participants with Best Response of CR or PR | Baseline up to approximately 4 years
  Per investigator assessed RECIST 1.1
Phase 1a and 1b-Time to Response (TTR) | Baseline up to approximately 4 years
  Per investigator assessed RECIST 1.1
Phase 1a and 1b-Progression-free Survival (PFS) | Baseline up to approximately 4 years
  Per investigator assessed RECIST 1.1
Phase 1a and 1b-Disease Control Rate (DCR) | Baseline up to approximately 4 years
  Per investigator assessed RECIST 1.1
Phase 1a and 1b-Duration of Response (DOR) | Baseline up to approximately 4 years
  Per investigator assessed RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (24):
- United States (15):
  - Stanford Cancer Center, Stanford, California
  - Florida Cancer Specialists - Lake Nona - Sarah Cannon Research Institute, Orlando, Florida
  - Florida Cancer Specialists - Sarasota, Sarasota, Florida
  - The University of Chicago Medical Center (UCMC), Chicago, Illinois
  - Community Health Network, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - John Theurer Cancer Center At Hackensack UMC, Hackensack, New Jersey
  - Columbia University, New York, New York
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - The Ohio State University (OSU) Wexner Medical Center, Columbus, Ohio
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - START Mountain Region, West Valley City, Utah
  - NEXT Virginia, Fairfax, Virginia
- France (2):
  - Centre Leon Berard, Lyon
  - Institut Gustave Roussy, Villejuif
- Japan (3):
  - Kyoto University Hospital, Kyoto
  - National Cancer Center Hospital, Tokyo
  - Cancer Institute Hospital of JFCR, Tokyo
- South Korea (2):
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Spain (2):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY4175408 in Participants With Advanced Cancer — https://trials.lilly.com/en-US/trial/624057